CLINICAL TRIAL: NCT06163079
Title: Assisted Reproductive Techniques (ART) With Sperm Donation : an Inclusive Model of ART for All Women
Acronym: PMAPT
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Mikael AGOPIANTZ, MCU-PH - ART Center coordinator, Central Hospital, Nancy, France
Other Study IDs: 2023PI128
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Fertility Issues
Keywords: parenthood; Assisted reproductive techniques
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Single women applying for sperm donation: Inclusion of all single women consulting the Reproductive Medicine Service for a parenthood project by sperm donation between January 2021 and June 2023.
  Exclusion :
  * Minors
  * Person under guardianship
  Interventions: Behavioral: No intervention
- women in relationship with a women applying for sperm donation: Inclusion of all women in relationship with a women consulting the Reproductive Medicine Service for a parenthood project by sperm donation between January 2021 and June 2023.
  Exclusion :
  * Minors
  * Person under guardianship
  Interventions: Behavioral: No intervention
- Heterosexuel couples applying for sperm donation: Inclusion of all heterosexual couples consulting the Reproductive Medicine Service for a parenthood project by sperm donation between January 2021 and June 2023.
  Exclusion :
  * Minors
  * Person under guardianship

INTERVENTIONS:
Behavioral: No intervention — No intervention. This is a retrospective study. Data will be collected from routine consultations Will be collectad the following datas : Number and evolution of requests, age, background, infertility timing, parenthood context, Appointment time, ART timing, Type of ART, ART outcome, Outcome time
  Groups: Single women applying for sperm donation; women in relationship with a women applying for sperm donation

SUMMARY:
This is a monocentric, retrospective, non-interventional study. The main objective is to describe the populations requesting assisted reproductive techniques (ART) with sperm donation ; and compare them between groups depending on their parental project..

The secondary objectives are to describe the center support process in the context of ART with sperm donation, to determine the initial/final orientation of support and the time to care The statistical analysis will be carried out to compare these parameters between groups depending on their parental project The study is taking place in the reproductive medicine department of the regional university hospital centre in Nancy.

DETAILED DESCRIPTION:
Descriptive analysis of a new MAP population since the update of bioethics legislation in August 2021 This study is a descriptive analysis of the population requesting assisted reproductive techniques (ART) with sperm donation since update of bioethics legislation in August 2021 ; and compare them in groups depending on their parental project.

The main objective is to describe the different populations requesting ART with sperm donation (number and evolution of requests, age, history, geographical origin, infertility delay, parenthood context).

The secondary objectives are to describe the center support process in the context of ART with sperm donation, to determine the initial/final orientation of support and the time to care and compare them between groups depending on their parental project

The statistical analysis will be carried out to compare these parameters between groups depending on their parental project

This research contributes to our knowledge of patients with a parental project. It may lead to improve their medical care

The study is monocentric, retrospective, non-interventional and does not involve human subjects. This research is based on existing data, extracted from patient files in the médifirst software.

This is taking place in the reproductive medicine department of the regional university hospital centre in Nancy.

ELIGIBILITY:
Inclusion Criteria:

* single women consulting the Reproductive Medicine Service for a parenthood project by sperm donation between January 2021 and June 2023.
* women in relationship with women consulting the Reproductive Medicine Service for a parenthood project by sperm donation between January 2021 and June 2023

Exclusion Criteria:

* Minors
* Person under guardianship

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: single women and women in relationship with women consulting the Reproductive Medicine Service for a parenthood project through sperm donation between January 2021 and June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
significant result p < 0.05 of qualitative and quantitative data | Statistical analysis will be performed by January 2024
  The significance of statistical tests (significant result p < 0.05) will show if a difference exists among people applying for sperm donation between single women, women in relationship with a women, compared with heterosexual couples.
  Qualitative data are available in the medical files created during the usual appointments in the Reproductive Medicine Department.

SECONDARY OUTCOMES:
ART process | Statistical analysis will be performed by January 2024
  Describe the support process in the context of ART with sperm donation Determine the initial/final orientation of support and the different timeframes for care.

CONTACTS AND LOCATIONS:
Overall Officials: AGOPIANTZ Mikael, PhD, Principal Investigator — Central HNF Nancy Regional University Hospital
Locations (1):
- Centre AMP Maternité Régionale de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No